CLINICAL TRIAL: NCT00002583
Title: A Phase III Prospective Randomized Study of Adjuvant Chemotherapy With Vinorelbine and Cisplatin in Completely Resected Non-Small Cell Lung Cancer With Companion Tumour Marker Evaluation
Brief Title: Vinorelbine + Cisplatin or No Further Therapy in Non-small Cell Lung Cancer That Has Been Surgically Removed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Eastern Cooperative Oncology Group (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR10; CAN-NCIC-BR10 (Other: PDQ); CLB-9795 (Other: CALGB); E-JBR10 (Other: ECOG); SWOG-JBR10 (Other: SWOG); GW-565/040; NCI-V94-0492 (Other Grant/Funding Number: NCI); CDR0000063698 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Observation (No Intervention): Observation only
- Chemotherapy (Active Comparator): Cisplatin and Vinorelbine
  Interventions: Drug: cisplatin; Drug: vinorelbine ditartrate

INTERVENTIONS:
Drug: cisplatin — 50 mg/m2 IV
  Arms: Chemotherapy
Drug: vinorelbine ditartrate — 25 mg/m2 IV
  Arms: Chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if combination chemotherapy is more effective than no further treatment for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of vinorelbine plus cisplatin with that of no further therapy in treating patients who have stage I or stage II non-small cell lung cancer that has been completely removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the duration of overall and disease-free survival in patients with completely resected non-small cell lung cancer (NSCLC) randomized to adjuvant chemotherapy with vinorelbine and cisplatin versus observation only. II. Confirm the prognostic significance of ras mutations when present in the primary tumor. III. Provide a comprehensive tumor bank linked to a clinical database for the further study of molecular markers in resected NSCLC. IV. Measure and compare the health-related quality of life of patients on both treatment arms. V. Evaluate any toxicity related to this treatment regimen.

OUTLINE: This is a randomized study. Patients are stratified according to participating institution, nodal status (N0 vs N1), and ras mutation status of primary tumor (absent vs present vs unknown). Patients are randomized to one of two treatment arms. Arm I: Patients are evaluated at 3 and 6 months after randomization. Arm II: Patients receive vinorelbine IV over 6-10 minutes weekly for 16 weeks. Patients also receive cisplatin IV on days 1 and 8 every 4 weeks for a total of 4 courses. Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at Canadian centers. Quality of life assessments are optional for ECOG and SWOG centers. Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 450 patients will be accrued for this study within 6.75 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary non-small cell lung cancer that is completely resected No mixed small and non-small cell histologies Pathologic T2 N0 or T1-2 N1 T1 N1 and T2 N1 only for CALGB institutions Removal of all gross disease with negative resection margins by lobectomy, sleeve resection, bilobectomy, or pneumonectomy (based on intraoperative findings) No segmentectomy or wedge resection Complete mediastinal lymph node resection or sampling required at primary tumor resection, with minimum levels of nodal sampling as follows: Primary in right upper lobe - levels 4, 7, 10 Primary in right middle lobe - levels 4, 7, 10 Primary in right lower lobe - levels 4, 7, 9, 10 Primary in left upper lobe - levels 5, 6, 7, 10 Primary in left lower lobe - levels 7, 9, 10 If complete mediastinal lymph node resection has not been undertaken, any mediastinal lymph node which measured 1.5 cm or more on presurgical CT scan must have been biopsied and found to be free of metastatic involvement Disease at nodal station 10 (tracheobronchial angle) is considered N2 disease for this trial and is not eligible No more than one discrete primary tumor No bronchoalveolar carcinoma with lobar or multilobar involvement Discrete solitary radiological mass or nodule eligible Snap frozen fresh primary tumor tissue must be submitted to Lung Cancer Tumor Bank within 14 days after surgery by selected Canadian centers Others to submit representative paraffin block within 2 months of surgery

PATIENT CHARACTERISTICS: Age: 18 and over (lower age limit determined by individual center) Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count greater than 2,000/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 10.0 g/dL Hepatic: Bilirubin no greater than 1.25 times normal AST/ALT no greater than 1.25 times normal Alkaline phosphatase no greater than 1.25 times normal Renal: Creatinine no greater than 1.7 mg/dL Cardiovascular: No history of congestive heart failure or other cardiac abnormality that may preclude hydration necessary for cisplatin administration Other: No active pathologic condition that would preclude study No active uncontrolled infection No history of psychiatric or neurologic disorder that would preclude study No prior breast cancer, melanoma, or hypernephroma No other malignancy within the past 5 years except adequately treated nonmelanomatous skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception Ability to tolerate treatment (based on consultation between the thoracic surgeon and a medical oncologist or hematologist) and available for follow-up

PRIOR CONCURRENT THERAPY: Complete resection required Randomization between 28 and 40 days after surgery required

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 1994-07-07 (Actual); Primary Completion 2004-04-25 (Actual); Study Completion 2009-12-21 (Actual)

PRIMARY OUTCOMES:
survival | At time of death

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L. Winton, MD, Study Chair — University of Alberta; Eric Vallieres, MD, FRCSC, Study Chair — University of Washington; Russell F. DeVore, MD, Study Chair — Vanderbilt-Ingram Cancer Center; James R. Rigas, MD, Study Chair — Norris Cotton Cancer Center
Locations (155):
- United States (135):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - University of Missouri, Columbia, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
- Canada (20):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - St. Paul's Hospital - Vancouver, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Hotel Dieu Hospital - St. Catharines, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asmis TR, Ding K, Seymour L, Shepherd FA, Leighl NB, Winton TL, Whitehead M, Spaans JN, Graham BC, Goss GD; National Cancer Institute of Canada Clinical Trials Group. Age and comorbidity as independent prognostic factors in the treatment of non small-cell lung cancer: a review of National Cancer Institute of Canada Clinical Trials Group trials. J Clin Oncol. 2008 Jan 1;26(1):54-9. doi: 10.1200/JCO.2007.12.8322. PMID 18165640
- [Background] Wheatley-Price P, Le Maître A, Ding K, et al.: The influence of sex on efficacy, toxicity and delivery of treatment in National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) non-small cell lung cancer (NSCLC) chemotherapy trials. [Abstract] J Clin Oncol 26 (Suppl 15): A-8054, 2008.
- [Background] Hicks L, Cheung M, Hasan B, et al.: Venous thromboembolism and non-small cell lung cancer: a pooled analysis of National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) trials. [Abstract] Blood 110 (11): A-3995, 2007.
- [Background] Kassam F, Shepherd FA, Johnston M, Visbal A, Feld R, Darling G, Keshavjee S, Pierre A, Waddell T, Leighl NB. Referral patterns for adjuvant chemotherapy in patients with completely resected non-small cell lung cancer. J Thorac Oncol. 2007 Jan;2(1):39-43. doi: 10.1097/JTO.0b013e31802baff6. PMID 17410008
- [Background] Ng R, Hasan B, Mittmann N, Florescu M, Shepherd FA, Ding K, Butts CA, Cormier Y, Darling G, Goss GD, Inculet R, Seymour L, Winton TL, Evans WK, Leighl NB; Working Group on Economic Analysis; Lung Disease Site Group; National Cancer Institute of Canada Clinical Trials Group. Economic analysis of NCIC CTG JBR.10: a randomized trial of adjuvant vinorelbine plus cisplatin compared with observation in early stage non-small-cell lung cancer--a report of the Working Group on Economic Analysis, and the Lung Disease Site Group, National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 Jun 1;25(16):2256-61. doi: 10.1200/JCO.2006.09.4342. PMID 17538170
- [Background] Hotta K, Matsuo K, Kiura K, Ueoka H, Tanimoto M. Advances in our understanding of postoperative adjuvant chemotherapy in resectable non-small-cell lung cancer. Curr Opin Oncol. 2006 Mar;18(2):144-50. doi: 10.1097/01.cco.0000208787.91947.a2. PMID 16462183
- [Background] Pignon JP, Tribodet H, Scagliotti GV, et al.: Lung Adjuvant Cisplatin Evaluation (LACE): a pooled analysis of five randomized clinical trials including 4,584 patients. [Abstract] J Clin Oncol 24 (Suppl 18): A-7008, 2006.
- [Background] Wakelee HA, Schiller JH, Gandara DR. Current status of adjuvant chemotherapy for stage IB non-small-cell lung cancer: implications for the New Intergroup Trial. Clin Lung Cancer. 2006 Jul;8(1):18-21. doi: 10.3816/CLC.2006.n.028. PMID 16870041
- [Background] Visbal AL, Leighl NB, Feld R, Shepherd FA. Adjuvant Chemotherapy for Early-Stage Non-small Cell Lung Cancer. Chest. 2005 Oct;128(4):2933-43. doi: 10.1378/chest.128.4.2933. PMID 16236970
- [Result] Butts CA, Ding K, Seymour L, Twumasi-Ankrah P, Graham B, Gandara D, Johnson DH, Kesler KA, Green M, Vincent M, Cormier Y, Goss G, Findlay B, Johnston M, Tsao MS, Shepherd FA. Randomized phase III trial of vinorelbine plus cisplatin compared with observation in completely resected stage IB and II non-small-cell lung cancer: updated survival analysis of JBR-10. J Clin Oncol. 2010 Jan 1;28(1):29-34. doi: 10.1200/JCO.2009.24.0333. Epub 2009 Nov 23. PMID 19933915
- [Result] Bezjak A, Lee CW, Ding K, Brundage M, Winton T, Graham B, Whitehead M, Johnson DH, Livingston RB, Seymour L, Shepherd FA. Quality-of-life outcomes for adjuvant chemotherapy in early-stage non-small-cell lung cancer: results from a randomized trial, JBR.10. J Clin Oncol. 2008 Nov 1;26(31):5052-9. doi: 10.1200/JCO.2007.12.6094. Epub 2008 Sep 22. PMID 18809617
- [Result] Jang RW, Le Maître A, Ding K, et al.: A Q-TWiST analysis of adjuvant chemotherapy in non-small cell lung cancer (NSCLC) in the NCIC CTG JBR.10 trial. [Abstract] J Clin Oncol 26 (Suppl 15): A-6535, 2008.
- [Result] Tsao MS, Zhu C, Ding K, et al.: A 15-gene expression signature prognostic for survival and predictive for adjuvant chemotherapy benefit in JBR.10 patients. [Abstract] J Clin Oncol 26 (Suppl 15): A-7510, 2008.
- [Result] Bezjak A, Lee CW, Ding K, et al.: Quality of life (QOL) impact of adjuvant chemotherapy for early stage non-small cell lung cancer (NSCLC): final analysis of JBR.10 randomized trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-7585, 405s, 2007.
- [Result] Gauthier I, Ding K, Winton T, Shepherd FA, Livingston R, Johnson DH, Rigas JR, Whitehead M, Graham B, Seymour L. Impact of hemoglobin levels on outcomes of adjuvant chemotherapy in resected non-small cell lung cancer: the JBR.10 trial experience. Lung Cancer. 2007 Mar;55(3):357-63. doi: 10.1016/j.lungcan.2006.10.021. Epub 2006 Dec 1. PMID 17141357
- [Result] Pepe C, Hasan B, Winton TL, Seymour L, Graham B, Livingston RB, Johnson DH, Rigas JR, Ding K, Shepherd FA; National Cancer Institute of Canada and Intergroup Study JBR.10. Adjuvant vinorelbine and cisplatin in elderly patients: National Cancer Institute of Canada and Intergroup Study JBR.10. J Clin Oncol. 2007 Apr 20;25(12):1553-61. doi: 10.1200/JCO.2006.09.5570. PMID 17442999
- [Result] Seve P, Lai R, Ding K, Winton T, Butts C, Mackey J, Dumontet C, Dabbagh L, Aviel-Ronen S, Seymour L, Whitehead M, Tsao MS, Shepherd FA, Reiman T. Class III beta-tubulin expression and benefit from adjuvant cisplatin/vinorelbine chemotherapy in operable non-small cell lung cancer: analysis of NCIC JBR.10. Clin Cancer Res. 2007 Feb 1;13(3):994-9. doi: 10.1158/1078-0432.CCR-06-1503. PMID 17289895
- [Result] Tsao MS, Aviel-Ronen S, Ding K, et al.: P53 protein over-expression but not p53 gene mutation is a poor prognostic marker and a predictive marker for survival benefit from adjuvant chemotherapy in non-small cell lung cancer (NSCLC) in the JBR.10 trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-7577, 403s, 2007.
- [Result] Pepe C, Hasan B, Winton T, et al.: Adjuvant chemotherapy in elderly patients: an analysis of National Cancer Institute of Canada Clinical Trials Group and Intergroup BR.10. [Abstract] J Clin Oncol 24 (Suppl 18): A-7009, 2006.
- [Result] Reiman T, Lai R, Ding K, et al.: Class III beta tubulin expression and benefit from adjuvant cisplatin/vinorelbine chemotherapy in operable non-small cell lung cancer: analysis of the National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) study JBR.10. [Abstract] J Clin Oncol 24 (Suppl 18): A-7051, 376s, 2006.
- [Result] Alam N, Shepherd FA, Winton T, Graham B, Johnson D, Livingston R, Rigas J, Whitehead M, Ding K, Seymour L. Compliance with post-operative adjuvant chemotherapy in non-small cell lung cancer. An analysis of National Cancer Institute of Canada and intergroup trial JBR.10 and a review of the literature. Lung Cancer. 2005 Mar;47(3):385-94. doi: 10.1016/j.lungcan.2004.08.016. PMID 15713522
- [Result] Gauthier I, Ding K, Winton T, et al.: Impact of hemoglobin (Hb) on outcomes of adjuvant chemotherapy (ACT) with cisplatin/vinorelbine in patients (pts) with completely resected non small cell lung cancer (NSCLC) in JBR.10. [Abstract] J Clin Oncol 23 (Suppl 16): A-7200, 670s, 2005.
- [Result] Winton T, Livingston R, Johnson D, Rigas J, Johnston M, Butts C, Cormier Y, Goss G, Inculet R, Vallieres E, Fry W, Bethune D, Ayoub J, Ding K, Seymour L, Graham B, Tsao MS, Gandara D, Kesler K, Demmy T, Shepherd F; National Cancer Institute of Canada Clinical Trials Group; National Cancer Institute of the United States Intergroup JBR.10 Trial Investigators. Vinorelbine plus cisplatin vs. observation in resected non-small-cell lung cancer. N Engl J Med. 2005 Jun 23;352(25):2589-97. doi: 10.1056/NEJMoa043623. PMID 15972865
- [Result] Winton TL, Livingston R, Johnson D, et al.: A prospective randomised trial of adjuvant vinorelbine (VIN) and cisplatin (CIS) in completely resected stage 1B and II non small cell lung cancer (NSCLC) Intergroup JBR.10. [Abstract] J Clin Oncol 22 (Suppl 14): A-7018, 621s, 2004.
- [Result] Alam N, Shepherd F, Winton T, et al.: Compliance with adjuvant chemotherapy (ACT) in non-small lung cancer (NSCLC): NCIC-CTG BR.10/JBR.10. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2547, 633, 2003.
- [Result] Beziak A, Winton T, Ding K, et al.: Quality of life in a trial of adjuvant chemotherapy for early stage completely resected non-small cell lung cancer (NCIC CTG BR.10). [Abstract] Lung Cancer 41 (Suppl 2): S20, 2003.